CLINICAL TRIAL: NCT05131841
Title: A Multi-center, Randomized, Open-label Study on Pharmacokinetics, Safety, Efficacy, and Immunogenicity of Cipterbin Combined With Vinorelbine Injection Every Week or Every Three Weeks in the Treatment of Patients With HER2-positive Metastatic Breast Cancer
Brief Title: Cipterbin Combined With Vinorelbine in the Treatment of HER2-positive MBC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Proswell Medical Corporation (Industry)
Responsible Party: Principal Investigator, wangxiaojia, Director, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-302H-mBC-IIT-01
Record Dates: First submitted 2021-09-03; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; HER2-positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-week group (Active Comparator): Cipterbin combined with Vinorelbine Injection every week in the treatment of patients with HER2-positive metastatic breast cancer
  Interventions: Drug: Cipterbin Combined With Vinorelbine
- Three-week group (Experimental): Cipterbin combined with Vinorelbine Injection every three weeks in the treatment of patients with HER2-positive metastatic breast cancer
  Interventions: Drug: Cipterbin Combined With Vinorelbine

INTERVENTIONS:
Drug: Cipterbin Combined With Vinorelbine — 1. Cipterbin combined with Vinorelbine Injection every week in the treatment of patients with HER2-positive metastatic breast cancer
  2. Cipterbin combined with Vinorelbine Injection every three weeks in the treatment of patients with HER2-positive metastatic breast cancer

SUMMARY:
To compare pharmacokinetics Index of Cipterbin combined with Vinorelbine Injection every week or every three weeks in the treatment of patients with HER2-positive metastatic breast cancer

DETAILED DESCRIPTION:
A multi-center, randomized, open-label study on pharmacokinetics, safety, efficacy, and immunogenicity of Cipterbin combined with Vinorelbine Injection every week or every three weeks in the treatment of patients with HER2-positive metastatic breast cancer. The main purpose was to compare pharmacokinetics Index between two groups, secondly to observe safety, efficacy, and immunogenicity

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤70 years old, female.
* BMI index in the range of 19.0~28.0
* ECOG≤1, and the expected os ≥3 months
* Unresectable metastatic breast cancer diagnosed by histology or pathology that has received one or more chemotherapy regimens.
* HER2 overexpression is +++ by immunohistochemistry (IHC) or + by fluorescence hybridization FISH.
* At least one measurable lesion.
* Sufficient organ function
* Voluntarily signed an informed consent form.
* Subjects with good compliance

Exclusion Criteria:

* Rapid disease progression or threaten important organs and require urgent replacement therapy.
* Undergone surgery within 28 days before treatment (except for biopsy)
* Received radiotherapy within 21 days before the first study drug treatment or the side effects of radiotherapy have not recovered to 0 or 1
* Suffer from other serious uncontrolled diseases (such as epilepsy, liver failure, kidney failure, etc.)
* Suffered from other malignant tumors within 5 years before receiving the first study drug treatment or at the same time.
* Severely infected
* Clear history of mental illness, or have a history of alcoholism or drug abuse.
* Central nervous system metastasis or meningeal metastasis with clinical symptoms
* Cardiac function left ventricular ejection fraction < 50%
* Obvious arrhythmia, myocardial ischemia, severe atrioventricular block, cardiac insufficiency, severe heart valve Membrane disease patients
* Poorly controlled hypertension
* Patients with coagulopathy: INR or APTT ≥1.5×ULN
* Allergic to the test drug or its excipients in the study treatment, or have a severe allergic reaction to other monoclonal antibody drugs in the past
* Pregnant or breastfeeding, or cannot take reliable contraceptive measures during the trial and within 6 months after the end of the medication Giver
* Have received a certain test drug in other interventional clinical trials, the interval is less than 28 days or less than 5 half lives of the drug (whichever is longer)
* Have used a monoclonal antibody within 6 months before receiving the first study drug treatment
* Have received other drugs that may affect the pharmacokinetic results of the study drug, the interval is less than 28 days or less than 5 half lives of the drug (whichever is longer)
* Have received organ transplants (including autologous/allologous stem cell transplants) in the past
* Other conditions judged by the investigator to be inappropriate for participating in this trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | From enrollment to 21 days after the last dose administrate
  Cmax after the last administration
Cmin | From enrollment to 21 days after the last dose administrate
  Cmin after the last administration
AUC0-t | From enrollment to 21 days after the last dose administrate
  AUC0-t after the last administration
AUCtau | From enrollment to 21 days after the last dose administrate
  AUCtau after the last administration

SECONDARY OUTCOMES:
Multiple sets of Cmax | From enrollment to 21 days after the last dose administrate
  Cmax after the first administration and the third administration in the three-week administration group and the seventh administration in the one-week administration group.
Multiple sets of Cmin | From enrollment to 21 days after the last dose administrate
  Cmin after the first administration and the third administration in the three-week administration group and the seventh administration in the one-week administration group.
Multiple sets of AUC0-t | From enrollment to 21 days after the last dose administrate
  AUC0-t after the first administration and the third administration in the three-week administration group and the seventh administration in the one-week administration group.
Multiple sets of AUCtau | From enrollment to 21 days after the last dose administrate
  AUCtau after the first administration and the third administration in the three-week administration group and the seventh administration in the one-week administration group.
Multiple sets of Tmax | From enrollment to 21 days after the last dose administrate
  Tmax after the first administration and the third administration in the three-week administration group and the seventh administration in the one-week administration group.
Safety index | From enrollment to 30 days after the last dose administrate
  Adverse Events during the test
BOR | From enrollment to death(for any reason),Until 24 months after the last subject left the administration group
  Record the proportion of CR and PR in all subjects
DCR | From enrollment to death(for any reason),Until 24 months after the last subject left the administration group
  CR/PR/SD accounted for the proportion of all subjects
OS | From enrollment to death(for any reason),Until 24 months after the last subject left the administration group
  Overall Survival of all subjects
Immunogenicity index | From enrollment to 21 days after the last dose administrate
  ADA

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, chief doctor, Study Director — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared from the trial begin for 10 years
Supporting Information: CSR
Time Frame: From the trial begin for 10 years
Access Criteria: Every one